CLINICAL TRIAL: NCT06101888
Title: A Prospective, Multicenter, Single-group Clinical Study to Evaluate the Safety and Efficacy of Peijia Medical Transcatheter Aortic Valve System in the Treatment of Severe Aortic Valve Regurgitation
Brief Title: Safety and Effectiveness of TaurusTrio™ Heart Valve System in Patients With Severe Aortic Regurgitation (AR)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peijia Medical Technology (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15CSP001
Record Dates: First submitted 2023-10-20; First posted 2023-10-26 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Aortic Regurgitation
MeSH Terms: conditions — Aortic Valve Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A single set of test (Experimental): The experimental apparatus consisted of TaurusTrio™ Heart Valve (THV), Delivery Catheter & Introducer Sheath ,Loading Tools
  Interventions: Device: TaurusTrio™ Heart Valve System

INTERVENTIONS:
Device: TaurusTrio™ Heart Valve System — The TaurusTrio™ Heart Valve System contains the following sub-components: a prosthetic transcatheter porcine pericardial aortic valve, 20Fr Introducer Sheath System, transfemoral Delivery Catheter, and Loading Tool.

SUMMARY:
To evaluate the safety and effectiveness of the TaurusTrio™ Heart Valve System in a patient population with symptomatic severe AR requiring replacement/repair of their native aortic valve that are at high risk for open surgical aortic valve replacement/repair (SAVR).

ELIGIBILITY:
Inclusion Criteria:

* Patients who voluntarily participate and sign the informed consent and are able to comply with the entire trial process;
* Age ≥ 18 years;
* Adult subjects with severe AR (Grade ≥ 3) as assessed by echocardiography based on ASE (American Society of Echocardiography) using multiparametric approach with:

  * Jet width ≥ 65% of LVOT
  * Vena contracta width of > 6 mm
  * Holodiastolic flow reversal in proximal abdominal/descending aorta
  * Jet deceleration rate/Pressure half time <200ms
  * AND, For Grade 3:
  * Regurgitant volume ≥ 45-59 ml/beat
  * Regurgitant fraction ≥ 40-49%
  * EROA ≥ 0.2-0.29 cm2
  * OR, For Grade 4:
  * Regurgitant volume ≥ 60 ml/beat
  * Regurgitant fraction≥50%
  * EROA ≥ 0.3 cm2 Note: In cases where not all criteria listed for severe AR are met, the Core Lab will determine severity. Supplemental CMR imaging may be used to substantiate the degree of AR reported by Core Lab on baseline echo when imaging is suboptimal, Doppler parameters are discordant or inconclusive regarding the severity of AR, or when a discrepancy is present between the echo findings and the clinical setting.
* Patients who have symptoms obviously caused by Aortic Regurgitation, such as dyspnea, chest pain, NYHA Class II or higher;
* Patients who are unsuitable for conventional surgery but needs TAVR（It is recommended to refer to the 2020 ACC/AHA Heart Valve Disease Management Guidelines when evaluating the risks of surgical valve surgery），evaluated by the cardiac team (including at least one interventional cardiologist and one cardiovascular surgeon)
* Patient has suitable anatomy to accommodate the insertion and delivery of the JenaValve Trilogy™ Heart Valve System，evaluated by core laboratory;

Exclusion Criteria:

* Congenital uni- or bicuspid aortic valve morphology；
* Previous prosthetic aortic valve (bioprosthesis or mechanical) implant；
* Mitral regurgitation or Tricuspid regurgitation> moderate；
* Clinically significant coronary artery disease (CAD) requiring revascularization within 30 days prior to index procedure, or planned CAD revascularization procedure within 12 months after index procedure；
* Echocardiographic evidence of left ventricular thrombus；
* Endocarditis within 180 days prior to index procedure；
* Hypertrophic cardiomyopathy with or without obstruction；
* Severe pulmonary hypertension (systolic PA pressure >80 mmHg)；
* Severe RV dysfunction as assessed clinically and by echo；
* Severely reduced left ventricular ejection fraction (LVEF <25%)；
* Aortic annular perimeter derived diameter of <21.0 mm or > 28.6 mm or perimeter <66.0 mm or >90 mm (assessed by Multi-Detector CT measurement)；
* Aortic annulus angulation > 70° (assessed by Multi-Detector CT measurement)；
* Straight length of ascending aorta of < 55 mm；
* Significant disease of ascending aorta, including ascending aortic aneurysm ； (defined as maximal luminal diameter of 50 mm or greater) or atheroma (including if thick [>5 mm], protruding or ulcerated)
* Need for urgent or emergent TAVR procedure for any reason；
* Cardiogenic shock or hemodynamic instability requiring inotropic support or ventricular assist device within 30 days prior to index procedure；
* Myocardial infarction < 30 days prior to index procedure；
* Cerebrovascular event (TIA, stroke) < 180 days prior to index procedure；
* Patients with common carotid artery or internal carotid artery or vertebral artery stenosis (>70%)；
* Patients with severe coagulopathy；
* Severe renal insufficiency (GFR < 30 ml/min) at Screening, OR renal disease requiring renal replacement therapy within 180 days prior to index procedure；
* Blood dyscrasias as defined: leukopenia (WBC < 3000/mm³), or thrombocytopenia (platelets < 90,000/µl) or anemia (Men: Hgb < 8.1 g/dl; Women: Hgb < 7.4 g/dl)；
* Active peptic ulcer or upper gastrointestinal bleeding < 90 days prior to index procedure；
* Known allergies to to heparin, aspirin, ticlopidine, Clopidogrel, Nitroglycerin and other drugs，contrast agents, nitinol shape memory alloy, tantalum or porcine products；
* Contraindication to intraoperative transesophageal echocardiography and/or Multi-Detector CT (MDCT) scan；
* Estimated life-expectancy of < 24 months；
* Patient is enrolled in another investigational medical device or drug study which has not completed the required primary endpoint follow-up. (Note: Patients involved in a long-term surveillance phase of another study are eligible for enrollment in this study);
* Other medical, social, or psychological conditions that in the opinion of an Investigator precludes the patient from providing appropriate informed consent;
* Severe dementia (resulting in either inability to provide informed consent for the trial/procedure, prevents independent lifestyle outside of a chronic care facility, or will fundamentally complicate rehabilitation from the procedure or compliance with follow-up assessments);
* Unable to comply with follow-up requirements;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality at 12 months | 12 months
  All-cause mortality

SECONDARY OUTCOMES:
Improvement in quality of life (QoL) at 12 months over baseline, as measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ). | 12 months
  Improvement in quality of life (QoL)
Composite safety endpoint at 30 days | 30 days after procedure
  all-cause death；all stroke； life-threatening or major bleeding；acute kidney injury (AKI) stage 2, 3 or dialysis；major vascular complications；surgery/intervention related to the device (including coronary intervention)；permanent pacemaker implantation；moderate or severe total aortic regurgitation

OTHER OUTCOMES:
Technical Success at exit from OR, hybrid room or cath lab post-index procedure | Immediate after procedure
  Absence of procedural mortality; and Successful access, delivery, and retrieval of transcatheter delivery system; and Deployment and correct positioning of a single intended THV; and Freedom from re-intervention related to the device or access procedure
Device Success at 1-month consisting of | 30 days after procedure
  Absence of procedure mortality; and Correct position of a single prosthetic heart valve Intended performance of the prosthetic heart valve (i.e., no prosthesis mismatch and mean aortic valve gradient <20 mmHg or peak velocity <3 m/s; and no moderate or severe prosthetic valve regurgitation) Intended performance of the prosthetic heart valve (i.e., no prosthesis mismatch and mean aortic valve gradient <20 mmHg or peak velocity <3 m/s; and no moderate or severe prosthetic valve regurgitation)
Procedural Success at 1-month consisting of | 30 days after procedure
  Device success at 30 days; and No device- or procedure-related serious adverse events (defined as below):
  i) No disabling or non-disabling stroke ii) No life-threatening bleeding (>4 units PRBC) iii) No acute kidney injury - Stage 2 or 3 (including dialysis) iv) No major vascular complication v) No myocardial infarction or cardiac ischemia requiring PCI or CABG vi) No valve-related dysfunction requiring repeat procedure (BAV, TAVI, or SAVR)

CONTACTS AND LOCATIONS:
Locations (19):
- China (19):
  - Beijing Anzhen Hospital, Beijing, Beijing Municipality
  - Fu Wai Hospital, Beijing, China, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - XiaMen Cardiovascular Hospital XiaMen University, Xiamen, Fujian
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangdong, Guangzhou
  - The Second Affiliated Hospital of Harbin Medical University, Haerbin, Heilongjiang
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Wuhan Union Hospital, China, Wuhan, Hubei
  - Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Nanjing First Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Namchang Umiversity, Nanchang, Jiangxi
  - General Hospital of Northern Theater Command, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Xijing Hospital, Xian, Shanxi
  - West China Hospital, Chengdu, Sichuan
  - Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital of Zhejiang, Hangzhou, Zhejiang